CLINICAL TRIAL: NCT06255054
Title: Novel Approaches to Assessing Cannabis Impaired Driving
Brief Title: Novel Approaches to Assessing Cannabis Impaired Driving (NAACID)
Acronym: NAACID
Status: Recruiting | Type: Observational
Sponsor: Colorado School of Public Health (Other)
Responsible Party: Principal Investigator, Ashley Brooks-Russell, Associate Professor, Director (Injury and Violence Prevention Center), Colorado School of Public Health
Other Study IDs: ColoradoSPH
Record Dates: First submitted 2023-07-21; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Cannabis Use
Keywords: Driving Impairment

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood specimens may be stored long-term with participant consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Non-Users: People who do not use cannabis.
- Daily Flower Users: People who use cannabis flower daily.
- Daily Concentrate Users: People who use cannabis concentrate products daily.
- Occasional Flower Users: People who use cannabis flower at least once a month and no more than three times per week.

SUMMARY:
Researchers at the University of Colorado Anschutz Medical Campus, Colorado School of Public Health, and Injury & Violence Prevention Center want to learn more about how people are affected by cannabis in different ways. We will use a driving simulator to compare the driving performance of adults who use cannabis daily, occasionally or have not recently used cannabis.

ELIGIBILITY:
Inclusion Criteria:

* The following are inclusion criteria for participants to be enrolled in any of the four phases of the study:

  1. Participants who are ≥21 years old and ≤55 years old
  2. Participants who are able to provide written, informed consent
  3. Participants with active healthcare coverage (including health insurance, Medicaid, etc.)
  4. Participants who are willing to complete up to two in-person study visits (one for Phases 1 & 2, and two for Phases 3 & 4), including up to two urine drug screens, two alcohol breathalyzer tests, and one urine pregnancy test (if applicable)
  5. Participants who agree to refrain from using non-prescription psychotropic drugs (e.g., ecstasy), hallucinogens, and synthetic cannabinoids during the study
  6. Participants who agree to refrain from drinking >3 alcoholic drinks the day prior to the data collection study visit (the single visit for Phases 1 & 2, and the second visit for Phases 3 & 4)
  7. Participants who agree to refrain from using any cannabis products for at least 8 hours prior to the data collection study visit (the single visit for Phases 1 & 2, and the second visit for Phases 3 & 4)
  8. Participants who are willing to provide and use their own cannabis product that has been procured from a licensed dispensary, is labeled with THC potency, and contains <2% CBD (cannabis use groups only; the single visit for Phases 1 & 2, and the second visit for Phases 3 & 4)
  9. Participants who agree to have a sober driver pick them up after the data collection study visit (cannabis use groups only; the single visit for Phases 1 & 2, and the second visit for Phases 3 & 4)
  10. Participants who take at least 2 inhalations ("hits") during their typical inhalational (smoking/vaporizing) sessions, or ingest at least 5 mg of THC when they consume edible cannabis products (cannabis use groups only)
  11. Participants who are willing to provide a sample of their cannabis to be independently tested for potency and terpene content (Phases 1, 3 & 4 only)

Exclusion Criteria:

* The following are exclusion criteria for participants to be enrolled in any of the four phases of the study:

  1. Prisoners
  2. Participants who have nocturnal schedules (e.g., work night shifts)
  3. Participants with a history of abuse or addiction to substances other than cannabis (e.g., prescription and non-prescription pharmaceuticals, alcohol, or illicit drugs)
  4. Participants who have expressed an interest in substance abuse treatment within the 60 days prior to study enrollment
  5. Participants who report consuming an average of >3 alcoholic drinks per day in the 30 days prior to study enrollment
  6. Participants with any past or current diagnosis of schizophrenia, narcolepsy, heart disease, epilepsy, or a traumatic brain injury
  7. Participants who are currently experiencing untreated bipolar disorder, major depression, sleep apnea, or other uncontrolled medical conditions as determined by the investigators (e.g., hypertension)
  8. Participants with a known balance or gait disorder
  9. Participants with color blindness (Phase 2 only)
  10. Participants who currently wear hard contact lenses for vision correction (Phase 2 only)
  11. Participants who have donated 450 mL or more of blood in the two weeks prior to study enrollment
  12. Participants who are pregnant or breastfeeding (female participants only)
  13. Participants who report never using cannabis before in their lifetime (Phases 1 & 2 only)
  14. Participants with a history of clinically significant adverse event(s) associated with cannabis intoxication (e.g., lightheadedness, nausea, dizziness, etc., cannabis use groups only)
  15. Participants with uncorrected visual acuity disorder, defined as binocular vision worse than 20/40 (Phases 2, 3 & 4 only; determined at screening)
  16. Participants with a body mass index >40 kg/m2 (determined at screening)
  17. Participants with a positive breath alcohol test (breathalyzer) at screening
  18. Participants who are otherwise unsuitable for inclusion in the study, based on the opinion of the investigator

Ages: 25 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: Potential participants will be recruited from the general population.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2020-06-20 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Driving Impairment | 5 years
  SDLP (standard deviation of lateral position) is measured by our Advanced NADS minisim

CONTACTS AND LOCATIONS:
Locations (1):
- Driving Study Lab, Denver, Colorado, United States